CLINICAL TRIAL: NCT03122587
Title: Non-Invasive Brain Stimulation and Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16-2342
Record Dates: First submitted 2017-04-04; First posted 2017-04-21 (Actual); Results first posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2019-07

CONDITIONS: Substance Use Disorders
Keywords: tACS; Brain Stimulation; Transcranial Alternating Current Stimulation; Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Active Sham (Session 1 and Session 2) (Sham Comparator): Active sham transcranial alternating current stimulation (tACS) during Session 1 and Session 2
  Interventions: Device: Active sham transcranial alternating current stimulation
- Active Sham (Session 1) and tACS at 10 Hz (Session 2) (Experimental): Active sham transcranial alternating current stimulation (tACS) during Session 1 and Transcranial Alternating Current Stimulation at 10 Hz during Session 2
  Interventions: Device: Transcranial Alternating Current Stimulation at 10 Hz
- Active Sham (Session 1) and tACS at 40 Hz (Session 2) (Experimental): Active sham transcranial alternating current stimulation (tACS) during Session 1 and Transcranial Alternating Current Stimulation at 40 Hz during Session 2
  Interventions: Device: Transcranial Alternating Current Stimulation at 40 Hz

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation at 10 Hz — Non-invasive, safe transcranial alternating current stimulation administered at 10 Hz to target alpha oscillatory activity
  Other Names: tACS at 10 Hz
  Arms: Active Sham (Session 1) and tACS at 10 Hz (Session 2)
Device: Transcranial Alternating Current Stimulation at 40 Hz — Non-invasive, safe transcranial alternating current stimulation administered at 40 Hz to target gamma oscillatory activity
  Other Names: tACS at 40 Hz
  Arms: Active Sham (Session 1) and tACS at 40 Hz (Session 2)
Device: Active sham transcranial alternating current stimulation — Active sham (placebo)
  Other Names: Active sham
  Arms: Active Sham (Session 1 and Session 2)

SUMMARY:
The will investigate the feasibility and effectiveness and initial efficacy of non-invasive transcranial alternating current stimulation (tACS) on distress tolerance and inhibitory control among treatment seeking substance users.

DETAILED DESCRIPTION:
Disruptions in inhibitory control (IC) and distress tolerance (DT) are implicated in the development and maintenance of substance use disorders. Findings suggest that differential DLPFC engagement during affective and cognitive processing, and in particular, distress tolerance, in substance use disorder may be malleable, providing a promising intervention. Modulating neural oscillations with non-invasive, safe brain stimulation by targeting regions such as the DLPFC may provide an avenue to improve distress tolerance and inhibitory control in SUD. Transcranial alternating current stimulation (tACS) may be a particularly promising approach as it is a safe and non-invasive method of electric stimulation that has the potential to effectively modulate neural network and circuit dynamics, more closely aligning with a network-based conceptualization of affective and cognitive processesThis study will test the effects of tACS on distress tolerance and inhibitory control among treatment-seeking adults with substance use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Current Diagnostic and Statistical Manual of Mental Disorders (DSM-V) Substance Use Disorder
* Current smoker
* Abstinent from all substances (except nicotine) for at least the past 2 weeks

Exclusion Criteria:

* Current use of antiepileptic drugs and/or benzodiazepines
* Less than 6 months since an electroconvulsive therapy (ECT) session
* Current DSM-V Psychotic Disorder
* Pregnancy and/or nursing
* Ongoing or history of traumatic brain injury (TBI), reoccurring seizures, stroke, or brain tumors
* Medical or neurological illness
* Brain devices and/or implants

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey B Daughters, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Southlight Healthcare, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Sham Stimulation (Session 1 and Session 2): Active sham transcranial alternating current stimulation: Active sham (placebo)
- Active Sham (Session 1) and tACS at 10 Hz (Session 2): Active Sham during Session 1 and Transcranial Alternating Current Stimulation at 10 Hz during Session 2
  Transcranial Alternating Current Stimulation at 10 Hz: Non-invasive, safe transcranial alternating current stimulation administered at 10 Hz to target alpha oscillatory activity
- Active Sham (Session 1) and tACS at 40 Hz (Session 2): Active Sham during Session 1 and Transcranial Alternating Current Stimulation at 40 Hz during Session 2
  Transcranial Alternating Current Stimulation at 40 Hz: Non-invasive, safe transcranial alternating current stimulation administered at 40 Hz to target gamma oscillatory activity
Period: Overall Study
Arm/Group | Active Sham Stimulation (Session 1 and Session 2) | Active Sham (Session 1) and tACS at 10 Hz (Session 2) | Active Sham (Session 1) and tACS at 40 Hz (Session 2)
Started | 13 | 12 | 13
Completed | 11 | 10 | 12
Not Completed | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Sham Stimulation (Session 1 and Session 2) | Active Sham (Session 1) and tACS at 10 Hz (Session 2) | Active Sham (Session 1) and tACS at 40 Hz (Session 2) | Total
Number analyzed (Participants) | 13 | 12 | 13 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (6.5) | 43.3 (9.5) | 42.9 (7.8) | 43.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 5 | 13
  Male | 8 | 9 | 8 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 5 | 11
  White | 7 | 8 | 7 | 22
  More than one race | 3 | 1 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 12 | 13 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change in Distress Tolerance (Mean Latency to Quit the PASAT-C)
Description: The Computerized Paced Auditory Serial Addition Task (PASAT-C) is a psychological distress-inducing task. Numbers are presented sequentially on a computer screen and participants are asked to add the currently presented number to the previously presented number before the next number is presented. Participants select the answer using a computer mouse on a number pad displayed on the computer screen below the presented numbers. The speed of the number presentations is individually titrated in order to account for some individual differences in cognitive capacity, but not to secure equal performance among individuals. Incorrect or delayed responses are met with an aversive explosion sound. Distress tolerance is the latency to task termination (i.e., time until quit in minutes).
Time Frame: From Session 1 to Session 2, up to 6 days
Population: 3 participants did not have data due to impedance issues, behavioral noncompliance, and technology error
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Active Sham Stimulation (Session 1 and Session 2) | Active Sham (Session 1) and tACS at 10 Hz (Session 2) | Active Sham (Session 1) and tACS at 40 Hz (Session 2)
Number analyzed (Participants) | 10 | 10 | 10
minutes | 11.2 (5.5) | 9.8 (6.4) | 9.4 (6.2)

2. Primary Outcome: Change in Inhibitory Control (Mean D-prime on the Go/No-Go)
Description: During the computerized Go/No-Go task, participants view a serial stream of pictures and are instructed to continuously press a button on the computer keyboard, but inhibit responses when stimuli are presented consecutively. Inhibitory control will be calculated as d-prime [z(hit rate) - z(false alarm rate)]. Each z-score of 0 is equal to the mean of the reference population, with a standard deviation of 1. Positive d-prime values indicate more inhibitory control, and negative values indicate less inhibitory control.
Time Frame: From Session 1 to Session 2, up to 6 days
Population: 3 participants did not have data due to impedance issues, behavioral noncompliance, and technology error
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Active Sham Stimulation (Session 1 and Session 2) | Active Sham (Session 1) and tACS at 10 Hz (Session 2) | Active Sham (Session 1) and tACS at 40 Hz (Session 2)
Number analyzed (Participants) | 10 | 10 | 10
z-score | -0.6 (2.0) | 0.9 (1.7) | -0.3 (1.9)

ADVERSE EVENTS:
Time Frame: From Session 1 to Session 2, up to 6 days
Groups:
- Active Sham Stimulation: Active sham transcranial alternating current stimulation: Active sham (placebo)
Arm/Group | Active Sham Stimulation | Active Sham (Session 1) and tACS at 10 Hz (Session 2) | Active Sham (Session 1) and tACS at 40 Hz (Session 2)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT03122587/Prot_SAP_000.pdf